CLINICAL TRIAL: NCT00728780
Title: Study to Compare the Bioavailability of ABT-335 and Rosuvastatin From ABT-143 Capsules Relative to That From Co-administration of ABT-335 and Rosuvastatin for the 5/45mg Dosage Form.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M10-586
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Adverse Events; Pharmacokinetic Variables
Keywords: Adverse events; Pharmacokinetic variables
MeSH Terms: interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): ABT-143 15/135mg
  Interventions: Drug: ABT-143
- B (Active Comparator): ABT-335 135mg and rosuvastatin 15mg
  Interventions: Drug: ABT-335 and rosuvastatin

INTERVENTIONS:
Drug: ABT-143 — once
  Arms: A
Drug: ABT-335 and rosuvastatin — once
  Arms: B

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of ABT-335 and rosuvastatin from ABT-143 relative to that from the co-administration of ABT-335 and rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Condition of good health

Exclusion Criteria:

* Currently enrolled in another study
* Females who are pregnant or breast feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Adverse events and safety laboratory assessments | 7 days
Pharmacokinetic parameters | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, Study Director — AstraZeneca
Locations (1):
- Site Reference ID/Investigator# 11101, Evansville, Indiana, United States